CLINICAL TRIAL: NCT01452178
Title: Observational Study on Peripheral Vascular Disease, Glucometabolic Status, and Type D Personality in Patients With Acute Myocardial Infarction.
Brief Title: Vastmanland Myocardial Infarction Study (VaMIS)
Acronym: VaMIS
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Västmanland County Council, Sweden (Other Government)
Responsible Party: Sponsor
Other Study IDs: VaMIS
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Acute Myocardial Infarction; Peripheral Artery Disease; Diabetes
Keywords: Cardiovascular diseases; Glucometabolic disorders; Type-D personality
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main purposes of this study are:

* to describe the prevalence of peripheral artery disease (including lower extremity artery disease, carotid artery disease, renal artery disease, and abdominal aortic disease) in patients with acute myocardial infarction in comparison to control subject from the general population,
* to evaluate the association of peripheral artery disease with glucometabolic status in patients with acute myocardial infarction,
* to assess the prevalence of type D personality in patients with acute myocardial infarction com pared to control subjects from the general population,
* to examine the prognostic value of peripheral artery disease in patients with acute myocardial infartion, and
* to evaluate the prognostic value of type D personality in patients with acute myocardial infarction.

DETAILED DESCRIPTION:
Atherosclerotic arterial disease is the main cause of premature death worldwide and is anticipated to remain the single leading cause of morbidity and mortality the following two decades. Coronary heart disease (CHD) and peripheral arterial disease (PAD) are important clinical manifestation of atherosclerosis which have common underlying arterial pathology, risk factors, and preventive treatments, but they are not often studied concurrently. In the view of secondary prevention we need to know more about the prevalence of cardiovascular disease and prognosis in patients at documented high risk, i.e. patients with manifested CHD. Previous studies on patients with CHD and concomitant PAD have focused mainly on either lower extremity PAD or carotid artery disease. In this project we expand the concept of PAD in patients with CHD to include lower extremity arterial disease, carotid artery disease, renal artery disease, and abdominal aortic aneurysmal disease.

Diabetes mellitus is a well recognised risk factor for cardiovascular morbidity and mortality. However, even prediabetic conditions carry an increased risk. One possible explanation for this increased risk may be the presence of a greater number of atherosclerotic lesions in patients with glucometabolic disorders than in patients without such disorders. We aim to evaluate the association of PAD with glucometabolic status in patients with manifest CHD.

A growing body of research has demonstrated the role of psychosocial and behavioural risk factors in the pathogenesis and prognosis of cardiovascular disorders. Recently, the type D ("distressed") personality construct has been proposed as a strong risk factor for cardiovascular morbidity and mortality. Type D personality is characterized by high levels of two personality traits: negative affectivity (e.g. worry, irritability, and gloom) and social inhibition (e.g. lack of self-assurance and reticence). The data on type D personality as a risk factor for cardiovascular disease has been limited to few research groups and there is a need to replicate those data in other populations.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at the Department of Cardiology, Central Hospital, Västerås, Sweden.
* Living in the catchment area of the Central Hospital, Västerås, Sweden.
* Diagnosis of acute myocardial infarction, i.e. a rise in serum concentration of troponin-I to >= 0.4 microgram/Liter and its subsequent fall in combination with one of the following: a) ischaemic symptoms, b) development of Q-waves on the ECG, c) ECG-changes indicative o ischaemia (ST segment elevation or depression), or d) coronary artery intervention.

Exclusion Criteria:

* age less than 18 years
* severly impaired communication capabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients hospitalized for acute myocardial infarction. Control subjects, matched to the patients for age, sex, and municipality, were randomly selected from the general population.
Sampling Method: Probability Sample
Enrollment: 1008 (Actual)
Dates: Start 2005-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of peripheral artery disease (lower extremity artery disease, carotid artery disease, renal artery disease, or abdominal aortic aneurysm) - cross sectional outcome measure. | baseline
  Peripheral artery disease as diagnosed by blood pressure measurements in ankles and arms (ankle-brachial-index) for lower extremity artery disease, or as diagnosed by ultrasonography for carotid artery disease, renal artery disease, or abdominal aortic aneurysm.
Prevalence of glucometabolic disorders - cross sectional outcome measure. | basline
  Known diabetes (from medical records), newly diagnosed diabetes, and impaired glucose tolerance (as diagnosed from plasma glucose levels and/or an oral glucose tolerance test.
Prevalence of type D personality - cross sectional measure. | baseline
  Type D personality as measured from the type D Scale-14 (DS14) questionnaire.
Cardiovascular events - longitudinal outcome measure. | 5-10 years
  Cardiovascular events obtained from the Swedish National Causes of Death register and the Swedish National In-Patient register. The registers are linked to the patients by the unique personal identification number assigned to each swedish resident.

CONTACTS AND LOCATIONS:
Overall Officials: Pär Hedberg, Assoc. Professor, Study Chair — Center for Clinical Research, Uppsala University, Västmanland County Hospital, SE-72189 Västerås, Sweden; Jerzy Leppert, Senior Professor, Principal Investigator — Center for Clinical Research, Uppsala University, Västmanland County Hospital, SE-72189 Västerås, Sweden
Locations (1):
- Center for Clinical Research, Uppsala University, Västmanland County Hospital, Västerås, Sweden

REFERENCES:
- [Result] Calais F, Frobert O, Rosenblad A, Hedberg PO, Wachtell K, Leppert J. Leisure-time physical inactivity and risk of myocardial infarction and all-cause mortality: a case-control study. Int J Cardiol. 2014 Dec 15;177(2):599-600. doi: 10.1016/j.ijcard.2014.08.137. Epub 2014 Aug 28. No abstract available. PMID 25223818
- [Result] Conden E, Rosenblad A, Ekselius L, Aslund C. Prevalence of type D personality and factorial and temporal stability of the DS14 after myocardial infarction in a Swedish population. Scand J Psychol. 2014 Dec;55(6):601-10. doi: 10.1111/sjop.12162. Epub 2014 Sep 22. PMID 25243796
- [Result] Selmeryd J, Henriksen E, Leppert J, Hedberg P. Interstudy heterogeneity of definitions of diastolic dysfunction severely affects reported prevalence. Eur Heart J Cardiovasc Imaging. 2016 Aug;17(8):892-9. doi: 10.1093/ehjci/jev211. Epub 2015 Sep 15. PMID 26374880
- [Result] Conden E, Rosenblad A. Insomnia predicts long-term all-cause mortality after acute myocardial infarction: A prospective cohort study. Int J Cardiol. 2016 Jul 15;215:217-22. doi: 10.1016/j.ijcard.2016.04.080. Epub 2016 Apr 15. PMID 27128534
- [Result] Hedberg P, Selmeryd J, Leppert J, Henriksen E. Long-term prognostic impact of left atrial volumes and emptying fraction in a community-based cohort. Heart. 2017 May;103(9):687-693. doi: 10.1136/heartjnl-2016-310242. Epub 2016 Nov 9. PMID 28067203
- [Result] Conden E, Rosenblad A, Wagner P, Leppert J, Ekselius L, Aslund C. Is type D personality an independent risk factor for recurrent myocardial infarction or all-cause mortality in post-acute myocardial infarction patients? Eur J Prev Cardiol. 2017 Mar;24(5):522-533. doi: 10.1177/2047487316687427. Epub 2017 Jan 10. PMID 28071958
- [Result] Eriksson Ostman M, Calais F, Rosenblad A, Frobert O, Leppert J, Hedberg P. Prognostic impact of subclinical or manifest extracoronary artery diseases after acute myocardial infarction. Atherosclerosis. 2017 Aug;263:53-59. doi: 10.1016/j.atherosclerosis.2017.05.027. Epub 2017 May 26. PMID 28599258
- [Result] Skau E, Henriksen E, Wagner P, Hedberg P, Siegbahn A, Leppert J. GDF-15 and TRAIL-R2 are powerful predictors of long-term mortality in patients with acute myocardial infarction. Eur J Prev Cardiol. 2017 Oct;24(15):1576-1583. doi: 10.1177/2047487317725017. Epub 2017 Aug 1. PMID 28762762
- [Result] Selmeryd J, Henriksen E, Dalen H, Hedberg P. Derivation and Evaluation of Age-Specific Multivariate Reference Regions to Aid in Identification of Abnormal Filling Patterns: The HUNT and VaMIS Studies. JACC Cardiovasc Imaging. 2018 Mar;11(3):400-408. doi: 10.1016/j.jcmg.2017.04.019. Epub 2017 Jul 19. PMID 28734926
- [Result] Calais F, Eriksson Ostman M, Hedberg P, Rosenblad A, Leppert J, Frobert O. Incremental prognostic value of coronary and systemic atherosclerosis after myocardial infarction. Int J Cardiol. 2018 Jun 15;261:6-11. doi: 10.1016/j.ijcard.2018.02.035. PMID 29657058
- [Result] Doerstling S, Hedberg P, Ohrvik J, Leppert J, Henriksen E. Growth differentiation factor 15 in a community-based sample: age-dependent reference limits and prognostic impact. Ups J Med Sci. 2018 Jun;123(2):86-93. doi: 10.1080/03009734.2018.1460427. Epub 2018 May 1. PMID 29714603
- [Result] Nilsson G, Hedberg P, Leppert J, Ohrvik J. Basic Anthropometric Measures in Acute Myocardial Infarction Patients and Individually Sex- and Age-Matched Controls from the General Population. J Obes. 2018 Oct 2;2018:3839482. doi: 10.1155/2018/3839482. eCollection 2018. PMID 30533220
- [Result] Nowak C, Carlsson AC, Ostgren CJ, Nystrom FH, Alam M, Feldreich T, Sundstrom J, Carrero JJ, Leppert J, Hedberg P, Henriksen E, Cordeiro AC, Giedraitis V, Lind L, Ingelsson E, Fall T, Arnlov J. Multiplex proteomics for prediction of major cardiovascular events in type 2 diabetes. Diabetologia. 2018 Aug;61(8):1748-1757. doi: 10.1007/s00125-018-4641-z. Epub 2018 May 24. PMID 29796748
- [Result] Henriksen E, Selmeryd J, Hedberg P. Associations of left atrial volumes and Doppler filling indices with left atrial function in acute myocardial infarction. Clin Physiol Funct Imaging. 2019 Jan;39(1):85-92. doi: 10.1111/cpf.12533. Epub 2018 Jul 1. PMID 29961999
- [Result] Velders MA, Calais F, Dahle N, Fall T, Hagstrom E, Leppert J, Nowak C, Tenerz A, Arnlov J, Hedberg P. Cathepsin D improves the prediction of undetected diabetes in patients with myocardial infarction. Ups J Med Sci. 2019 Aug;124(3):187-192. doi: 10.1080/03009734.2019.1650141. Epub 2019 Aug 20. PMID 31429631
- [Result] Cederlof ET, Johnston N, Leppert J, Hedberg P, Lindahl B, Christersson C. Do self-reported pregnancy complications add to risk evaluation in older women with established cardiovascular disease? BMC Womens Health. 2019 Dec 16;19(1):160. doi: 10.1186/s12905-019-0851-x. PMID 31842885
- [Result] Lodder P, Wicherts JM, Antens M, Albus C, Bessonov IS, Conden E, Dulfer K, Gostoli S, Grande G, Hedberg P, Herrmann-Lingen C, Jaarsma T, Koo M, Lin P, Lin TK, Meyer T, Pushkarev G, Rafanelli C, Raykh OI, Schaan de Quadros A, Schmidt M, Sumin AN, Utens EMWJ, van Veldhuisen DJ, Wang Y, Kupper N. Type D Personality as a Risk Factor for Adverse Outcome in Patients With Cardiovascular Disease: An Individual Patient-Data Meta-analysis. Psychosom Med. 2023 Feb-Mar 01;85(2):188-202. doi: 10.1097/PSY.0000000000001164. Epub 2023 Jan 9. PMID 36640440
- [Result] Nilsson G, Leppert J, Ohrvik J. Enigma of the cholesterol paradox in acute myocardial infarction: lessons from an 8-year follow-up of all-cause mortality in an age-matched and sex-matched case-control study with controls from the patients' recruitment area. BMJ Open. 2022 Jul 27;12(7):e057562. doi: 10.1136/bmjopen-2021-057562. PMID 35896296